CLINICAL TRIAL: NCT06336668
Title: Source of Human Milk Fortifier and Intestinal Oxygenation in Preterm Infants <30 Weeks Gestation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Belal Alshaikh, Principal Investigator, University of Calgary
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: REB23-1283
Record Dates: First submitted 2024-03-21; First posted 2024-03-29 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Feeding; Difficult, Newborn
Keywords: Feed intolerance; Human Milk fortifier; Bovine based Human Milk Fortifier; Human milk based Human Milk Fortifier; Preterm infants

STUDY DESIGN:
Intervention Model Description: Prospective randomized-controlled crossover trial comparing 2 different HMFs and 2 intestinal rSO2S periods in random order: 6 hours while on B-HMF and 6 hours on H-HMF with at least 6 hours washing period
Who Masked: Investigator
Masking Description: Randomizing the participants to either Bovine-HMF or Human Milk based-HMF will mask the Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bovine based-HMF (Active Comparator): The infant will fed human milk fortified with bovine-based HMF.
  Interventions: Dietary Supplement: Human milk-based HMF
- Human milk-based HMF (Experimental): The infant will be fed human milk fortified with human milk-based HMF.
  Interventions: Dietary Supplement: Human milk-based HMF

INTERVENTIONS:
Dietary Supplement: Human milk-based HMF — The study subject will be fed human milk fortified with a human-milk-based HMF.

SUMMARY:
Preterm infants require higher nutritional intakes during the neonatal phase than they do at any other stage of their development. Standard volumes of human milk alone do not offer sufficient nourishment to these infants. There are multiple options for fortifying human milk, which vary depending on whether the fortifier is derived from bovine sources (B-HMF) or human sources (H-HMF). Fortifying human milk has been proven to enhance growth in preterm infants without raising the risk of necrotizing enterocolitis (NEC), though it could potentially affect feeding tolerance. Changes in blood flow and oxygen levels in the intestines are commonly observed in infants experiencing feeding intolerance. Research indicates that feeding a mother's own milk (MOM) doesn't affect splanchnic (intestinal) oxygenation, whereas it decreases when feeding bovine-derived human milk fortifiers (B-HMF) or preterm formula, indicating greater oxygen requirements in the intestines of preterm infants fed these alternatives.

The goal of this clinical trial is to compare the effect of H-HMF and B-HMF on splanchnic oxygenation in infants less than 30 weeks.

DETAILED DESCRIPTION:
The fortification of human milk has been proven to enhance growth without raising the risk of necrotizing enterocolitis, although it may affect feeding tolerance.

Non-invasive techniques like Doppler ultrasonography of the superior mesenteric artery (SMA) and near-infrared spectroscopy (NIRS) have been utilized to evaluate mesenteric blood flow and intestinal oxygenation in preterm infants. Numerous studies have investigated the relationship between SMA flow and feeding intolerance. Findings indicate a significant correlation between increased mean Superior Mesenteric Artery blood flow velocity and early tolerance of enteral feeding. Moreover, research suggests a higher incidence of necrotizing enterocolitis (NEC) in preterm infants exhibiting increased resistance patterns of SMA blood flow velocity on the first day.

Non-invasive monitoring methods offer the ability to assess the impact of various fortification products on intestinal perfusion and oxygenation. This could aid in determining the most suitable fortification product to minimize episodes of feeding intolerance.

ELIGIBILITY:
Inclusion Criteria:

1. Preterm infants born <30 weeks' gestation age and less than 1500g of weight.
2. Admitted in Neonatal Intensive Care Unit at Foothills Medical Center
3. Reached full fortified enteral feed and at least 21 days of chronological age.

Exclusion Criteria:

1. Chromosomal or major congenital anomalies
2. Infants diagnosed with NEC.

Max Age: 30 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in Splanchnic regional oxygenation(rSO2S) measured by Near Infrared Spectroscopy | 6 hours
  Measurements of Near Infrared Spectroscopy are continuous but readings of interest are: before feeding, 30 and 120 minutes after finishing feed.

SECONDARY OUTCOMES:
Changes in SMA doppler peak flow velocity (PSV) | 6 hours
  SMA doppler will be performed before feed, and 30 and 120 minutes after completing the feed.
Changes in SMA doppler end-diastolic velocity (EDV) | 6 hours
  SMA doppler will be performed before feed, and 30 and 120 minutes after completing the feed.
Changes in SMA doppler Porcelout's resistance index (RI) | 6 hours
  SMA doppler will be performed before feed, and 30 and 120 minutes after completing the feed.

CONTACTS AND LOCATIONS:
Overall Officials: Belal Alshaikh, MD, MSCE, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No